CLINICAL TRIAL: NCT03638713
Title: Division of Gastroenterology, Department of Internal Medicine, Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Chiayi, Taiwan
Brief Title: Comparison of Procedural Sequences in Same-day Painless Bidirectional Endoscopy With Colonoscopic Water Exchange Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: A10604001
Record Dates: First submitted 2018-07-02; First posted 2018-08-20 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Colon Disease; Bidirectional Endoscopy
Keywords: water exchange; colonoscopy; cecal insertion time; bidirectional endoscopy
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Intervention Model Description: A total of 200 patients were allocated into one of two groups by computerized randomization. Patients in the group A (colonoscopy first group) received colonoscopy followed by EGD and those in the group B (EGD first group) received EGD followed by colonoscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- colonoscopy first group (Experimental): Patients received water-exchange colonoscopy first and followed by esophagogastroduodenoscopy
  Interventions: Behavioral: colonoscopy first
- EGD first group (Active Comparator): Patients received esophagogastroduodenoscopy first and followed by water-exchange colonoscopy
  Interventions: Behavioral: EGD first

INTERVENTIONS:
Behavioral: colonoscopy first — Received water exchange colonoscopy followed by EGD
  Arms: colonoscopy first group
Behavioral: EGD first — Received EGD followed by water exchange colonoscopy
  Arms: EGD first group

SUMMARY:
This prospective randomized controlled trial is to compare evaluate the optimal procedure sequence among patients undergoing water exchange colonoscopy.

DETAILED DESCRIPTION:
Same-day esophagogastroduodenoscopy (EGD) and colonoscopy (bidirectional endoscopy; BDE) are commonly performed to evaluate for gastrointestinal conditions, such as active gastrointestinal bleeding, iron deficiency anemia, positive fecal occult blood tests and abdominal pain. EGD-colonoscopy sequence seems to be the reasonable choice for BDE using air or CO2. With the use of water exchange method, endoscopists have to remove the dirty fecal material and air bubble during insertion. Gas insufflated during EGD may get into the colon and make subsequent water exchange colonoscopy more difficult. The aim of this prospective randomized controlled trial is to compare evaluate the optimal procedure sequence among patients undergoing water exchange colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent fully sedated bidirectional endoscopy in the physical check-up department

Exclusion Criteria:

* Patients who < 18 years old, > 80 years old
* Without standard colon preparation
* Allergy to meperidine or propofol
* With a history of partial colectomy
* Refusal to provide written informed consent
* American Society of Anesthesiology (ASA) risk Class 3 or higher

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
cecal insertion time | 30 minutes
  Cecal insertion time was defined as the time from insertion into the rectum to the time when the colonoscope tip passed to a point proximal to the ileocecal valve so that the base of cecum was visible.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsi Hsieh, MD, Study Director — Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Taipei, Taiwan

REFERENCES:
- [Derived] Hsieh YH, Koo M, Tseng CW. Comparison of Procedural Sequences in Sedated Same-Day Bidirectional Endoscopy with Water-Exchange Colonoscopy: A Randomized Controlled Trial. J Clin Med. 2022 Mar 2;11(5):1365. doi: 10.3390/jcm11051365. PMID 35268456